CLINICAL TRIAL: NCT02324387
Title: Assessment of the Tumor Response to Neoadjuvant Chemotherapy in Women With Locoregional Invasive Breast Cancer Using Tc99m Sestamibi Molecular Breast Imaging: A Prospective Study
Brief Title: Tc99m Sestamibi Molecular Breast Imaging
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014-0812; NCI-2015-00035 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2014-12-11; First posted 2014-12-24 (Estimated); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Molecular breast imaging; MBI; Tc99m sestamibi; Neoadjuvant chemotherapy; NAC
MeSH Terms: conditions — Breast Neoplasms | interventions — Technetium Tc 99m Sestamibi

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (1):
- Molecular Breast Imaging (MBI) + Tc99m sestamibi (Experimental): Participants undergo 3 MBI scans with injections of injection of Tc99m sestamibi before each scan. First scan is 7 days before scheduled chemotherapy treatment, after 2 cycles of chemotherapy, and after completion of chemotherapy treatment.
  Interventions: Procedure: Molecular Breast Imaging (MBI); Drug: Tc99m sestamibi

INTERVENTIONS:
Procedure: Molecular Breast Imaging (MBI) — Participants undergo 3 MBI scans with injections of injection of Tc99m sestamibi before each scan. First scan is 7 days before scheduled neoadjuvant chemotherapy (NAC) treatment, after 2 cycles of chemotherapy, and after completion of chemotherapy treatment.
  Other Names: MBI
Drug: Tc99m sestamibi — 8 mCi of 99mTc sestamibi by vein before each molecular breast imaging (MBI).

SUMMARY:
This clinical trial studies technetium Tc-99m sestamibi molecular breast imaging in predicting tumor response in patients with locoregional breast cancer that has spread from where it began in the breast to surrounding normal tissue who are receiving neoadjuvant chemotherapy. Comparing results of diagnostic procedures, such as technetium Tc-99m sestamibi molecular breast imaging, done before, during, and after chemotherapy may help doctors predict a patient's response to treatment and help plan the best treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the ability of technetium Tc-99m sestamibi (Tc 99m sestamibi) molecular breast imaging (MBI) to predict early response to neoadjuvant chemotherapy (NAC) and to assess residual disease at the completion of NAC in patients with locoregional invasive breast cancer.

SECONDARY OBJECTIVES:

I. To evaluate and qualitatively characterize Tc 99m sestamibi uptake by tumor on MBI at the baseline, after 2 cycles of NAC and at the completion of NAC.

II. To compare assessment of tumor response to NAC by MBI with digital mammography (DM), and breast ultrasound (US) exams.

III. To compare tumor size and distribution observed from MBI at the completion of NAC with extent of residual disease at surgery by pathological evaluation.

IV. To develop image acquisition and processing algorithm that quantifies the Tc 99m tumor uptake.

EXPLORATORY OBJECTIVE:

I. To determine effect of molecular subtype of cancer (Her2+, ER/PR/Her2- and ER+/Her2-) on diagnostic performance of MBI in predicting treatment response.

OUTLINE:

Patients undergo technetium Tc-99m sestamibi molecular breast imaging over 45 minutes at baseline (before start of NAC), after 2 courses of NAC (6-12 weeks, depending on the regimen), and the completion of NAC but before surgery. Patients also undergo breast ultrasound and mammographic imaging as standard of care at the same time points.

ELIGIBILITY:
Inclusion Criteria:

1. Female of 18 years and older of any race
2. Has biopsy-proven invasive breast cancer (BI-RADS 6) and scheduled for neoadjuvant chemotherapy (NAC).
3. Newly diagnosed biopsy proven locoregional invasive breast cancer at MD Anderson Cancer Center, or referred to MD Anderson for treatment after initial radiologic (mammographic, sonographic, etc.) exams at an outside institution in whom NAC is planned.
4. Patients with stage T1 or greater (T1-T4), nodal involvement (N0 - N3), without metastasis (M0) invasive breast cancer, including patients with inflammatory breast cancer.
5. Patients who agree to sign an informed consent to undergo MBI

Exclusion Criteria:

1. Is under 18 years of age
2. Is pregnant (confirmed by the patient as Imaging Clinic standard of care) or nursing mother
3. Has lesions involving chest wall
4. Has known allergy to Tc99m sestamibi

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2015-06-15 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Detection of Treatment Response using Molecular Breast Imaging (MBI) plus Tc99m sestamibi | 24 weeks
  Evaluation of treatment response by molecular breast imaging (MBI) tumor to background ratio (T/B), defined as T/B = ROIt_max/ROIb_mean, calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Gaiane M. Rauch, MD, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Lopez BP, Rauch GM, Adrada B, Kappadath SC. Functional tumor diameter measurement with molecular breast imaging: development and clinical application. Biomed Phys Eng Express. 2022 Aug 12;8(5). doi: 10.1088/2057-1976/ac85f0. PMID 35917778
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org